CLINICAL TRIAL: NCT01174537
Title: Clinical Application of Intravenous New Castle Disease Virus - HUJ Oncolytic Virus in the Treatment of Advanced Glioblastoma Multiforme, Soft and Bone Sarcomas and Neuroblastoma Patients, Resistant to Conventional Anti- Cancer Modalities
Brief Title: New Castle Disease Virus (NDV) in Glioblastoma Multiforme (GBM), Sarcoma and Neuroblastoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: ReuvenOr, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NDV-HUJ-HMO-CTIL
Record Dates: First submitted 2010-08-02; First posted 2010-08-03 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2010-08

CONDITIONS: Glioblastoma; Sarcoma; Neuroblastoma
Keywords: NDV; Metastatic; Refractory; Cancer; Progression-free; survival; recurrent
MeSH Terms: conditions — Glioblastoma; Sarcoma; Neuroblastoma; Neoplasm Metastasis; Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: New Castle Disease Virus — Patients will receive IV 1*10^10 EID50 (50 percent Embryo Infectious Dose. One EID50 unit is the amount of virus that will infect 50 percent of inoculated eggs) on a daily basis for a minimum of 5 days a week until disease progression for a minimum duration of 1 year.

SUMMARY:
Patients with specific metastatic cancers who failed prior therapeutic regimes will be treated with NDV for at least a year or until disease progression. The study will measure progression-free disease and posits that it will be extended.

DETAILED DESCRIPTION:
Present therapeutic regimes have not much improved the survival of patients with metastatic cancer. Therapeutic cancer vaccines are a form of immunotherapy designed to educate the immune system to recognise tumor cells as foreign rather than self. New Castle Virus (NDV) has a long history as a broad system oncolytic that can destroy tumor cells and stimulate the immune system. Up to 30 patients suffering from recurrent, refractory Glioblastoma Multiforme, soft an bone sarcomas and disseminated neuroblastoma will be enrolled in this trial and receive daily doses of NDV at least 5 days a week for a minimum of a year or until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of progressive disease in the above categories evaluated by standard tumor staging.
* Histologically confirmed diagnosis.
* Failure of conventional anti- cancer modalities.despite optimal application of all relevant available anti- cancer modalities.
* Age between 3 and 75 years old.
* Liver function tests less than twice the normal, renal function no more than 20% reduction and white cell and platelets count no more than 30% reduction.
* Karnofsky performance status of 50% or greater
* A written informed consent understood and signed by the patient and by a spouse, parent or guardian. In patients with GBM two signs will be required due to possible alterations of psych and understanding.

Exclusion Criteria:

* Not fulfilling any of the above criteria
* Moribund patients or patients with life- expectancy < 3 months
* Karnofksy performance status < 50%
* Pregnant or lactating women
* Active local or systemic infections requiring treatment
* Patients receiving other investigational agents
* History of allergy to egg ova-albumin.
* Co-morbidity or life- threatening clinical condition other than the basic cancer

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | at least 1 year
  Measure progression-free survival of patients receiving New Castle Virus

CONTACTS AND LOCATIONS:
Overall Officials: Reuven Or, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Gerl R, Vaux DL. Apoptosis in the development and treatment of cancer. Carcinogenesis. 2005 Feb;26(2):263-70. doi: 10.1093/carcin/bgh283. Epub 2004 Sep 16. PMID 15375012
- [Background] Zitvogel L, Apetoh L, Ghiringhelli F, Kroemer G. Immunological aspects of cancer chemotherapy. Nat Rev Immunol. 2008 Jan;8(1):59-73. doi: 10.1038/nri2216. PMID 18097448
- [Background] Ravindra PV, Tiwari AK, Sharma B, Chauhan RS. Newcastle disease virus as an oncolytic agent. Indian J Med Res. 2009 Nov;130(5):507-13. PMID 20090097
- [Background] Vigil A, Park MS, Martinez O, Chua MA, Xiao S, Cros JF, Martinez-Sobrido L, Woo SL, Garcia-Sastre A. Use of reverse genetics to enhance the oncolytic properties of Newcastle disease virus. Cancer Res. 2007 Sep 1;67(17):8285-92. doi: 10.1158/0008-5472.CAN-07-1025. PMID 17804743
- [Background] Freeman AI, Zakay-Rones Z, Gomori JM, Linetsky E, Rasooly L, Greenbaum E, Rozenman-Yair S, Panet A, Libson E, Irving CS, Galun E, Siegal T. Phase I/II trial of intravenous NDV-HUJ oncolytic virus in recurrent glioblastoma multiforme. Mol Ther. 2006 Jan;13(1):221-8. doi: 10.1016/j.ymthe.2005.08.016. Epub 2005 Oct 28. PMID 16257582
- [Background] Nelson NJ. Scientific interest in Newcastle disease virus is reviving. J Natl Cancer Inst. 1999 Oct 20;91(20):1708-10. doi: 10.1093/jnci/91.20.1708. No abstract available. PMID 10528013
- [Background] Schirrmacher V, Griesbach A, Ahlert T. Antitumor effects of Newcastle Disease Virus in vivo: local versus systemic effects. Int J Oncol. 2001 May;18(5):945-52. doi: 10.3892/ijo.18.5.945. PMID 11295039
- [Background] Lowe SW, Lin AW. Apoptosis in cancer. Carcinogenesis. 2000 Mar;21(3):485-95. doi: 10.1093/carcin/21.3.485. PMID 10688869